CLINICAL TRIAL: NCT03657472
Title: An Open-label, Randomized, Single-dose, 3-period Replicated Crossover Study to Compare the Pharmacokinetics and Safety Following Administration of CJ-30061 Alone and Co-administration of Amlodipine/Valsartan and Atorvastatin in Healthy Adult Volunteers
Brief Title: Bioequivalence Study of CJ-30061 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CJ_EXA_103
Record Dates: First submitted 2018-08-09; First posted 2018-09-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Hypertension; Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — Amlodipine, Valsartan Drug Combination; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sequence 1(RTR) (Experimental)
  Interventions: Drug: CJ-30061; Drug: Exforge® 5/160mg & Lipitor® 20mg
- Sequence 2(RRT) (Experimental)
  Interventions: Drug: CJ-30061; Drug: Exforge® 5/160mg & Lipitor® 20mg
- Sequence 3(TRR) (Experimental)
  Interventions: Drug: CJ-30061; Drug: Exforge® 5/160mg & Lipitor® 20mg

INTERVENTIONS:
Drug: CJ-30061 — Test: CJ-30061(Fixed-dose combination drug containing Amlodipine 5mg/Valsartan 160mg/Atorvastatin 20mg)
Drug: Exforge® 5/160mg & Lipitor® 20mg — Reference: Co-administration of Exforge® tab 5/160mg and Lipitor® tab 20mg

SUMMARY:
To compare the pharmacokinetics and safety after a single dose administration of CJ-30061 and co-administration of Exforge® 5/160mg, Lipitor® 20mg in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male aged 19 to 55 years at the time of signing informed consent form.
* Subject with BMI from 19kg/m^2 to 27kg/m^2
* Decided to participate in the study and provided signed informed consent form volutarily after receiving explanation of the objectives, contents, and property of Investigational products of the study

Exclusion Criteria:

* Subject who had a medical history of severe hepatobiliary, renal, gastrointestinal, cardiovascular, respiratory, endocrinological, neuropsychological, hematological, musculoskeletal disease.
* Subject who fall under the criteria below in laboratory test.

  * AST/ALT, total bilirubin, GGT, Uric acid > UNL (upper normal limit) x 1.5
  * CPK > UNL x 2.5
  * CrCL < 60mL/min
* Subject who fall under the criteria below in Blood Pressure test (siSBP < 100mmHg/siSBP ≥ 150mmHg or siDBP < 70mmHg/siDBP ≥ 100mmHg)

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2016-10-29 (Actual); Study Completion 2016-11-09 (Actual)

PRIMARY OUTCOMES:
Cmax of amlodipine | Up to 72 hours
Cmax of valsartan | Up to 72 hours
Cmax of atorvastatin | Up to 72 hours
AUCt of amlodipine | Up to 72 hours
AUCt of valsartan | Up to 72 hours
AUCt of atorvastatin | Up to 72 hours

SECONDARY OUTCOMES:
tmax of amlodipine | Up to 72 hours
tmax of valsartan | Up to 72 hours
tmax of atorvastatin | Up to 72 hours
t1/2 of atorvastatin | Up to 72 hours
t1/2 of amlodipine | Up to 72 hours
t1/2 of valsartan | Up to 72 hours
AUCinf of amlodipine | Up to 72 hours
AUCinf of valsartan | Up to 72 hours
AUCinf of atorvastatin | Up to 72 hours
AUCt of 2-OH atorvastatin | Up to 72 hours
Cmax of 2-OH atorvastatin | Up to 72 hours
tmax of 2-OH atorvastatin | Up to 72 hours
t1/2 of 2-OH atorvastatin | Up to 72 hours
AUCinf of 2-OH atorvastatin | Up to 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: JaeWook Ko, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No